CLINICAL TRIAL: NCT01062542
Title: Fertility in Female Cancer Survivors - Novel Assessment of Ovarian Reserve
Brief Title: Assessment of Ovarian Reserve in Female Cancer Survivors
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other); Canadian Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: UHN REB 08-0115-B
Record Dates: First submitted 2010-01-21; First posted 2010-02-04 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Breast Cancer Survivor; Pediatric Cancer Survivor
MeSH Terms: interventions — Blood Specimen Collection; High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Breast Cancer Survivors
  Interventions: Procedure: Blood Draw and Ultrasound
- Pediatric Cancer Survivors
  Interventions: Procedure: Blood Draw and Ultrasound
- Control group
  Interventions: Procedure: Blood Draw and Ultrasound

INTERVENTIONS:
Procedure: Blood Draw and Ultrasound — Patients will have a Blood sample taken to check hormone levels. Patients will also have an ultrasound test done to examine the ovaries. The ultrasound test is done by inserting a cylindrical probe into the vagina. The test has to be done this way to measures the ovaries accurately.

SUMMARY:
Chemotherapy can damage the ovaries and cause premature menopause. In women treated before the age of 40 years, menopause does not usually occur. We have very little information about the impact of chemotherapy on ovarian function in this particular group of women. In this study, we will check hormone blood tests and ultrasound tests of the ovaries to measure the reserve of eggs left in the ovaries after treatment in young survivors of breast cancer and childhood cancer. We will do the same tests in our comparison group. We can use these results to estimate the reduction in fertility in young cancer survivors.

DETAILED DESCRIPTION:
As women across North America and Europe increasingly delay childbirth, fertility preservation is emerging as an important issue among young breast cancer patients. The dramatic increase in survival for the major pediatric cancers in the last 50 years has resulted in an expanding population of childhood cancer survivors. The information currently available to counsel these patients about the impact of treatment on their fertility is inadequate. A significant degree of subfertility can exist prior to the onset of frank ovarian failure, and current studies do not address this.

This study will adopt new technologies that have revolutionized the evaluation of female fertility to assess ovarian function in young breast cancer survivors. The results will provide new, more accurate and clinically useful information to patients and physicians about the impact of cancer therapy on fertility. The results have the potential to influence clinical decisions regarding cancer treatment, and the use of assisted reproductive technologies for contemporary patients and survivors. Further, insofar as treatment advances are designed to improve disease control while reducing toxicity, these results may serve as the basis for better understanding the toxicity of modern therapy and provide opportunities for improvement.

ELIGIBILITY:
Inclusion Criteria:

* Breast Cancer Survivors

  1. histological confirmation of breast cancer
  2. received chemotherapy +/- radiotherapy with curative intent
  3. age 40 years or less at the time of diagnosis
  4. currently age 50 years or less
  5. currently disease free.
* Pediatric Cancer Survivors

  1. Received chemotherapy and / or radiotherapy with curative intent.
  2. Currently age 18 years and older.
  3. Currently premenopausal and attained at age 50 years or less.
  4. Currently disease free.
  5. Diagnosed with sarcoma or Hodgkin's disease or leukemia at 30 years or less.
* Control group 1. Premenopausal.

Exclusion Criteria:

* Breast Cancer Survivors

  1. treatment for malignancy other than breast cancer, involving chemotherapy or radiation to the ovaries/pelvis.
  2. any cancer recurrence
  3. hysterectomy/oophorectomy.
* Pediatric Cancer Survivors

  1. Hysterectomy / oophorectomy.
  2. Pelvic Radiation.
* Control group

  1. Received chemotherapy and / or pelvic radiation therapy,
  2. hysterectomy/oophorectomy.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients are selected from their primary care clinic.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2008-09; Primary Completion 2018-03 (Actual); Study Completion 2018-03-02 (Actual)

PRIMARY OUTCOMES:
To estimate the immediate decline in ovarian reserve in young breast cancer patients receiving chemotherapy using new biochemical and biophysical measures | 3 years
To model the decline in ovarian reserve with advancing age after cancer therapy in both young breast cancer and childhood cancer survivors and compare this with the decline seen in controls | 3 years
To develop methods to estimate the time to onset of menopause, and the time before natural or assisted conception such as in vitro fertilization become less successful | 3 years

SECONDARY OUTCOMES:
To evaluate the changes in ovarian function associated with specific chemotherapy regimens. | 3 years
To determine the time-to-pregnancy and cumulative incidence of pregnancy among young cancer survivors attempting pregnancy after treatment. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: David Hodgson, MD, Principal Investigator — University Health Network, Princess Margaret Hospital
Locations (1):
- University Health Network, Princess Margaret Hospital, Toronto, Ontario, Canada